CLINICAL TRIAL: NCT02872688
Title: A Baseline Controlled, Open Label, Single-arm Study to Investigate the Influence of GanedenBC30 (Bacillus Coagulans GBI-30, 6086) on the Gut Microbiome in Healthy Adults
Brief Title: Influence of GanedenBC30 (Bacillus Coagulans GBI-30, 6086) on the Gut Microbiome in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Collaborators: Ganeden Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GANERPD-160001-RPD01
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GanedenBC30 (Experimental)
  Interventions: Other: GanedenBC30

INTERVENTIONS:
Other: GanedenBC30
  Other Names: Bacillus coagulans GBI-30, 6086

SUMMARY:
The purpose of this study is to investigate the effect of a GanedenBC30, a probiotic bacteria (Bacillus coagulans strain GBI-30, 6086), on the gut microbiome in healthy adults. Subjects will complete a 2-week run-in period prior to receiving GanedenBC30. The study is open-label and subjects will act as their own controls as the microbiome is unique to individuals. During the run-in period, subjects will collect two stool samples and complete daily bowel habit diaries in order to understand usual habits and profile the microbiome for each subject. 30 subjects will take part in this research study conducted at Nutrasource Diagnostics Inc. Subjects will take GanedenBC30 for four weeks. Stool samples will be collected at the end of the study and daily bowel habit diaries maintained for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker, or ex-smoker ≥6 months
* Body mass index 18.5- 34.9 kg/m2 (inclusive)
* Female subjects of childbearing potential [i.e. not surgically sterilized or post-menopausal (greater than one year since last menses)] must have negative urine pregnancy test and must be using an effective birth control method
* Willing to avoid alcohol consumption for 24 h prior to every clinic visit
* Willing to maintain their regimens of dietary supplements known to alter GI function (including, but not limited to, iron supplements and calcium)
* Willing to maintain a stable body weight, activity level and dietary pattern except for use of the study products, as directed
* Willing and able to provide informed written consent

Exclusion Criteria:

* Pregnancy or lactation, or subject unwilling to take appropriate contraceptives for the duration of the study
* Use of prescription drugs (other than birth control) within 1 month prior to visit 1b
* Use of any weight-loss programs or weight-loss medications (prescription or over-the counter) including, but not limited to, lipase inhibitors, within 3 months prior to visit 1b
* Use of over-the-counter or prescription laxatives or stool softeners within 1 month prior to visit 1b
* Use of antibiotics (other than topical) within 2 months prior to visit 1b
* Use of prebiotic supplements (e.g. fructans and galacto-oligosaccharides (GOS), psyllium, fiber, inulin) or probiotic supplements (i.e. live microorganisms) within 1 month of visit 1b or consumption of any yogurts or foods with added prebiotics or added probiotics within 2 weeks of visit 1b
* History of blood clotting disorders or use of coagulation-inhibiting drugs (e.g. warfarin)
* Individuals with achlorhydria
* Presence of any disease (including, but not limited to: diabetes, gastrointestinal disease, cardiovascular disease, pancreatic, renal, or liver disease, chronic diarrhea or constipation, irritable bowel syndrome, or inflammatory bowel disease
* Abdominal or gastrointestinal surgery within the previous 12 months or planned abdominal or gastrointestinal surgery in the next 4 months
* Recent gastrointestinal food-borne illness (within 1 month prior to visit 1b)
* History of neurological disease (e.g. Parkinson's disease, stroke, traumatic brain injury, etc.)
* History of cancer (excluding non-melanoma skin cancer and basal cell carcinoma) in the past 5 years
* Controlled or uncontrolled hypertension defined as a seated resting systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
* Abnormal laboratory test results of clinical significance, including, but not limited to ALT or AST ≥1.5X the upper limit of normal at screening
* Presence or history (past 6 months) of alcohol or drug abuse; alcohol use of >2 standard alcoholic drinks per day
* Extreme dietary habits (e.g. vegan or very low carbohydrate diets)
* Subject has a known allergy or intolerance to soy
* Allergy or intolerance to or contraindication to both of the rescue antibiotic regimens (Ciprofloxacin and Septra (contains Trimethoprim)
* Subject is unwilling or unable to abide by the requirements of the protocol
* Any condition that would interfere with the subject's ability to comply with study instructions, might confound the interpretation of the study, or put the subject at risk
* Subject has taken an investigational health product or has participated in a research study within 30 days prior to first study visit

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12-19 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Changes in the gut microbiome | 4 weeks
  Observe changes in the gut microbiome after 4 weeks of supplementation with GanedenBC30 as assessed by 16s RNA sequencing of feces

SECONDARY OUTCOMES:
Change in stool frequency | 4 weeks
Change in stool consistency | 4 weeks
  Calculated using the Bristol stool scale form rating each bowel movement and averaging over each week
Changes severity of bloating as assessed by daily scores using a 4 point Likert scale | 4 weeks
  Determined using a 4 point Likert scale
Changes severity of gas as assessed by daily scores using a 4 point Likert scale | 4 weeks
Changes severity of abdominal pain as assessed by daily scores using a 4 point Likert scale | 4 weeks
Changes in feeling of overall well-being as assessed by daily scores using a 5 point Likert scale | 4 weeks

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by MedDRA coding | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource Diagnostics Inc., Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No